CLINICAL TRIAL: NCT02325076
Title: The Association Between Pulmonary Function Tests and Difficult Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Serkan Dogru, Assistant Professor, MD, Tokat Gaziosmanpasa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-KAEK-215
Record Dates: First submitted 2014-12-11; First posted 2014-12-24 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Airway Obstruction
Keywords: Airway Management; intubation; pulmonary function test
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spirodoc (Experimental): One time during examination at the outpatient unit
  Interventions: Device: Spirodoc

INTERVENTIONS:
Device: Spirodoc — A device to detect the physical condition of the lungs

SUMMARY:
The airflow moving from mouth to the lungs, which can be measured by pulmonary function tests, may be affected by the anatomic disorders of the upper airway. Difficult airway can be considered as the anatomic disorder of the upper airway as well. Therefore, there can be a relationship between difficult airway and pulmonary function tests. The purpose of this study is to elucidate the association between the pulmonary function tests and difficult airway.

DETAILED DESCRIPTION:
After approval of the Gaziosmanpasa University Clinical Trials Ethics Committee, patients those admitted to the anesthesiology outpatient unit will informed about the study. And pulmonary function tests by using Spirodoc® will be performed to those willing to participate in the study. Measurements of the pulmonary function tests, and measurements belong to difficult airway will be recorded.

In the operating theatre, after induction of anesthesia, the difficult intubation measurements will be recorded.

Normality and variance will be tested using One Sample Kolmogorov-Smirnov test, skewness, kurtosis and histograms for each variable. Quantitative data will present as means and standard deviation, and qualitative data as frequency and percentage. Depending on these results, Spearman's correlation analysis will perform to show the association between pulmonary function tests and difficult airway measurements. Analyses were conducted using the Statistical Package for Social Sciences program (SPSS Inc., Chicago, IL), version 20.0. Statistical significance for all analyses was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose admitted to the Gaziosmanpasa University, Medical Faculty, Anesthesiology and Reanimation outpatient unit
* Patients whose will be planned to undertake a surgical operation under general anesthesia and those performed tracheal intubation to secure the airway.
* An American Society of Anesthesiologists score of 1 or 2

Exclusion Criteria:

* Patient whose planned to undertake a surgical operation in the departments of ear-nose-throat, cardiac and vascular surgery, plastic and reconstructive surgery
* Patients with a history of chronic obstructive lung diseases
* Patients with a history of surgery on the neck
* Patients with a history of mandibular surgery

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Pulmonary function test differences between Mallampati 3 and 4 patients | eighteen months

SECONDARY OUTCOMES:
Cormack-Lehane grade | eighteen months
  Cormack-Lehane grade
Maximum mouth opening | eighteen months
  Maximum mouth opening
Percentage of glottic opening | eighteen months
  Percentage of glottic opening
Upper lip bite test score | eighteen months
  Upper lip bite test score
Measurement of neck circumference | eighteen months
  Measurement of neck circumference
Sterno-mental distance | eighteen months
  Sterno-mental distance
Thyromental distance | eighteen months
  Thyromental distance
Mean inspiratory flow | eighteen months
The ratio of forced expiratory flow 25% to forced expiratory flow 75% | eighteen months

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Dogru, Assist.Prof., Principal Investigator — Tokat Gaziosmanpasa University
Locations (1):
- Gaziosmanpasa University, Tokat Province, Tokat Province, Turkey (Türkiye)

REFERENCES:
- [Background] Leiter JC. Upper airway shape: Is it important in the pathogenesis of obstructive sleep apnea? Am J Respir Crit Care Med. 1996 Mar;153(3):894-8. doi: 10.1164/ajrccm.153.3.8630569.
- [Background] Tucker Woodson B. Structural effectiveness of pharyngeal sleep apnea surgery. Sleep Med Rev. 2008 Dec;12(6):463-79. doi: 10.1016/j.smrv.2008.07.010. PMID 19010290
- [Derived] Dogru S, Karaman T, Sahin A, Tapar H, Karaman S, Arici S, Suren M, Kaya Z, Somuk BT. Prediction of difficult laryngoscopy using spirometry: a pilot study. J Clin Monit Comput. 2017 Dec;31(6):1115-1121. doi: 10.1007/s10877-016-9961-2. Epub 2016 Nov 19. PMID 27866310